CLINICAL TRIAL: NCT06744985
Title: Mortality Prediction in Multiple Trauma Patients: A Comparison of the Revised Trauma Score and MGAP Score at a Trauma Center
Brief Title: Comparison of RTS and MGAP Scores in Predicting Outcomes of Trauma Patients
Acronym: RTS-MGAP
Status: Recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241213; 014 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-12; First posted 2024-12-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Multiple Trauma/Injuries
Keywords: RTS; MGAP
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this prospective cohort study is to compare the predictive accuracy of the Revised Trauma Score (RTS) and the MGAP score in determining clinical outcomes among multiple trauma patients hospitalized at a trauma center in Iraq.

The main questions it aims to answer are:

Which score, RTS or MGAP, provides a more accurate prediction of clinical outcomes, including mortality? Are there specific subgroups of trauma patients where one scoring system outperforms the other?

Participants will:

Be assessed using both the RTS and MGAP scores upon admission. Have their clinical outcomes, including mortality and other relevant indicators, monitored throughout their hospital stay.

DETAILED DESCRIPTION:
Trauma is one of the top four causes of mortality in developing countries and the second leading cause of death among the youth in these countries, as well as being the primary cause of year of life lost (YLL). Trauma represents a significant public health issue all over the world. With the progress of scientific and technological advancements and the industrialization of societies over the past century, trauma and its associated complications have emerged as the leading contributors to mortality and disability among individuals aged 1 to 44. Trauma represents a time-sensitive condition. Proper and effective management of trauma patients in both pre-hospital and hospital settings contributes to reducing mortality and preventing complications. The primary objectives in managing trauma patients include the rapid assessment of critically ill individuals, establishing treatment priorities, and delivering suitable care services.

Throughout the years, the rates of mortality due to trauma in Iraq have varied greatly because of different conflict-related influences. At the onset of the Iraq War in 2003, the case fatality rate (CFR) stood at approximately 20.4%, but by 2017 it had dropped to around 10.1%, indicating better survival outcomes among injured individuals. A study that examined combat-related fatalities from 2003 to 2006 found that although the monthly death count had doubled, the overall CFR stayed constant.

Scoring systems have been classically classified as anatomical, physiological, or combined scoring systems. The AIS, ISS, and NISS represent anatomical scoring systems that utilize various anatomical factors, such as the site and intensity of injuries. In contrast, the GCS, RTS, and PHI are physiological scoring systems that can be derived from data obtained during physical examinations. Additionally, the TRISS, NTRISS, and a TRISS are combined scoring systems that incorporate both anatomical and physiological characteristics of trauma.

The revised trauma score (RTS) is a physiological scoring system employed to assess trauma patients. Initially developed and assessed through a study involving over 2,000 individuals (10), the RTS incorporates three key physiological indicators: the Glasgow coma scale (GCS), systolic blood pressure (SBP), and respiration rate (RR). In addition, MGAP is primarily a physiological score that has been developed to predict survival outcomes in individuals experiencing trauma. Although it has been validated in research settings, it remains underutilized in low- and middle-income regions, despite its promise and practicality. The acronym MGAP represents the mechanism of injury (M), the Glasgow Coma Scale (G) score, the patient's age (A), and the systolic blood pressure (P). This score has previously been validated in France for its ability to predict 30-day mortality.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to the trauma center within 6 hours of injury.
* Availability of complete clinical and demographic data for scoring using RTS and MGAP.
* Patients who consent to participate in the study or whose legal representatives provide consent.
* Capability to assess outcomes such as survival, ICU admission, and complications.

Exclusion Criteria:

* Patients who expired before scoring or evaluation
* Missing or unreliable medical data for RTS or MGAP score calculations.
* Transfers from other facilities with interventions that could impact RTS or MGAP reliability.
* Pregnant patients, due to the unique considerations of trauma in pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multiple trauma patients were admitted to the trauma and emergency department at Al-Kadhimiya Teaching Hospital in Baghdad.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 7 days through discharge)
  Mortality (death) during hospitalization.
Accuracy Assessment of the Revised Trauma Score (RTS) | the first 6 hours after ER admission
  The total RTS score ranges from 0 to approximately 12, with lower scores indicating more severe injuries and a higher risk of mortality.
Accuracy Assessment of the MGAP score | the first 6 hours after ER admission
  (mechanism, Glasgow coma scale, age, and blood pressure), Total scores can range from 3 to 29, with a higher score predicting a better prognosis.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 7 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Number of Participants Requiring ICU Admission | Up to discharge, an average of 7 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Number of Participants Requiring Surgical Intervention | Up to discharge, an average of 7 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Bashar A Abdulhassan, Assistant professor of surgery, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly JF, Ritenour AE, McLaughlin DF, Bagg KA, Apodaca AN, Mallak CT, Pearse L, Lawnick MM, Champion HR, Wade CE, Holcomb JB. Injury severity and causes of death from Operation Iraqi Freedom and Operation Enduring Freedom: 2003-2004 versus 2006. J Trauma. 2008 Feb;64(2 Suppl):S21-6; discussion S26-7. doi: 10.1097/TA.0b013e318160b9fb. PMID 18376168
- [Background] Heydari Farhad. The effects of multidisciplinary education for nurses and physicians on the management of patients with multiple trauma.
- [Background] Heydari F, Maghami MH, Esmailian M, Zamani M. The Effect of Implementation of the Standard Clinical Practice Guideline (CPG) for Management of Multiple Trauma Patients Admitted to an Emergency Department. Adv J Emerg Med. 2017 Dec 11;2(1):e5. doi: 10.22114/AJEM.v0i0.37. eCollection 2018 Winter. PMID 31172068
- [Result] Sartorius D, Le Manach Y, David JS, Rancurel E, Smail N, Thicoipe M, Wiel E, Ricard-Hibon A, Berthier F, Gueugniaud PY, Riou B. Mechanism, glasgow coma scale, age, and arterial pressure (MGAP): a new simple prehospital triage score to predict mortality in trauma patients. Crit Care Med. 2010 Mar;38(3):831-7. doi: 10.1097/CCM.0b013e3181cc4a67. PMID 20068467
- [Result] Javali RH, Krishnamoorthy, Patil A, Srinivasarangan M, Suraj, Sriharsha. Comparison of Injury Severity Score, New Injury Severity Score, Revised Trauma Score and Trauma and Injury Severity Score for Mortality Prediction in Elderly Trauma Patients. Indian J Crit Care Med. 2019 Feb;23(2):73-77. doi: 10.5005/jp-journals-10071-23120. PMID 31086450
- [Result] Domingues CA, Coimbra R, Poggetti RS, Nogueira LS, de Sousa RMC. New Trauma and Injury Severity Score (TRISS) adjustments for survival prediction. World J Emerg Surg. 2018 Mar 6;13:12. doi: 10.1186/s13017-018-0171-8. eCollection 2018. PMID 29541155
- [Result] Soni KD, Mahindrakar S, Gupta A, Kumar S, Sagar S, Jhakal A. Comparison of ISS, NISS, and RTS score as predictor of mortality in pediatric fall. Burns Trauma. 2017 Aug 8;5:25. doi: 10.1186/s41038-017-0087-7. eCollection 2017. PMID 28795055
- [Result] Roy N, Gerdin M, Schneider E, Kizhakke Veetil DK, Khajanchi M, Kumar V, Saha ML, Dharap S, Gupta A, Tomson G, von Schreeb J. Validation of international trauma scoring systems in urban trauma centres in India. Injury. 2016 Nov;47(11):2459-2464. doi: 10.1016/j.injury.2016.09.027. Epub 2016 Sep 20. PMID 27667119
- [Result] Baghi I, Shokrgozar L, Herfatkar MR, Nezhad Ehsan K, Mohtasham Amiri Z. Mechanism of Injury, Glasgow Coma Scale, Age, and Systolic Blood Pressure: A New Trauma Scoring System to Predict Mortality in Trauma Patients. Trauma Mon. 2015 Aug;20(3):e24473. doi: 10.5812/traumamon.24473. Epub 2015 Aug 1. PMID 26543842
- [Result] Farzan N, Foroghi Ghomi SY, Mohammadi AR. A retrospective study on evaluating GAP, MGAP, RTS and ISS trauma scoring system for the prediction of mortality among multiple trauma patients. Ann Med Surg (Lond). 2022 Mar 28;76:103536. doi: 10.1016/j.amsu.2022.103536. eCollection 2022 Apr. PMID 35495411